CLINICAL TRIAL: NCT02800265
Title: A Pilot Study Evaluating the Bioavailability and Mucosal Bioactivity of the Dietary Supplement, Avmacol®, in Healthy Volunteers With Optimization of Buccal Cell Biomarkers
Brief Title: Bioavailability and Mucosal Bioactivity of Avmacol® in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Julie E. Bauman, MD, MPH, MD, MPH, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-204
Record Dates: First submitted 2016-06-02; First posted 2016-06-15 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: healthy volunteer; healthy; cancer prevention; prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avmacol during week 2 for 3 days (Experimental): Buccal cells line the inner cheek, and will be collected from the inner right cheek with a cytobrush (a q-tip like swab) by a trained investigator.
  During the second week the participant will take 8 Avmacol tablets every evening for 3 evenings (Day 2, 3, 4), and record the time of each dose in the provided diary. Research blood collection: on days 1 and 5. Overnight urine collection.
  Interventions: Dietary Supplement: Avmacol

INTERVENTIONS:
Dietary Supplement: Avmacol — Avmacol is an over-the-counter mixture of broccoli seed and sprout extracts in tablet form to promote detoxification. These tablets contain natural substances that stimulate the body's own defense mechanisms against toxic substances commonly encountered in the environment, such as air pollution and tobacco smoke.
  Other Names: Sulforaphane Production System; broccoli seed and sprout extract

SUMMARY:
Avmacol is an over-the-counter dietary supplement containing broccoli seed and sprout extracts in tablet form, hypothesized to activate protective cellular pathways including detoxication. In this study, healthy volunteers will take 3 days of Avmacol in order to evaluate both bioavailability and its bioactivity in cheek cells.

DETAILED DESCRIPTION:
Avmacol is an over-the counter dietary supplement containing broccoli seed and sprout extracts in tablet form. Natural plant substances within Avmacol, called phytochemicals, are hypothesized to stimulate the body's own defense mechanisms against toxic substances commonly encountered in the environment, such as air pollution and tobacco smoke. The purpose of this study is twofold: 1) to assess the protective effects of Avmacol on the mucosa (cheek cells) of healthy volunteers, and 2) to assess the collection of cheek cells by scraping, as a less invasive method of studying drug effects in the body compared to drawing blood or a tissue biopsy. Ultimately, these results will be used to design a larger study of Avmacol in patients with tobacco-related head and neck cancer. Avmacol will be studied as a way to possibly prevent a second cancer from developing in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Members of all racial and ethnic groups are eligible.
3. Smoking and non-smoking people are eligible. The tobacco use assessment form must be completed following consent and registration.
4. No chronic use of steroids
5. Karnofsky Performance Scale ≥90%
6. Able to provide written, informed consent
7. For women of child-bearing potential (WOCBP), a negative urine pregnancy test must be documented within 7 days prior to the first study intervention
8. Willing to avoid cruciferous vegetables during the study interventions
9. Willing to avoid grapefruit or grapefruit juice 48 hours prior to or during the study
10. Willing to avoid daily vitamins and anti-inflammatory medications prior to and during the study
11. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of study participation.
12. Willing and able to perform self-collection of buccal cells as stated in the instruction manual

Exclusion Criteria:

1. No current or former diagnosis of cancer, with the exception of: carcinoma-in-situ of breast or cervix; non-melanomatous skin cancer; T1-2, N0, M0 differentiated thyroid carcinoma; superficial bladder cancer; T1a or T1b prostate cancer comprising < 5% of resected tissue with normal prostate specific antigen (PSA) since resection
2. No use of chronic prescribed medications which are potent inducers or inhibitors of CYP3A4
3. Chronic use anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Number of buccal (cheek) cells collected by participants versus a trained professional | 5 days
  Number of buccal cells collected by cytobrush during week 1 (days 1-5) of the study

SECONDARY OUTCOMES:
Induction of NRF2 pathway transcripts in buccal cells by Avmacol | 5 days
  Quantitative mRNA for NQO1 in buccal cells at baseline (day 1) vs. buccal cells taken during the 3 days of Avmacol (days 2-4), and the day after Avmacol (day 5)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bauman, MD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No